CLINICAL TRIAL: NCT04110262
Title: Sodium Regulation in Individuals on Known Dietary Sodium Intake
Brief Title: Human Sodium Balance Study
Acronym: MEASURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Cheryl Anderson, Professor / Dean, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HL140488
Record Dates: First submitted 2019-08-23; First posted 2019-10-01 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
Keywords: Blood pressure; Sodium; Salt; Randomized controlled trial; balance; humans
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Dietary intervention consisting of two 25-day feeding periods separated by a 10-day washout.
Who Masked: Outcomes Assessor
Masking Description: Throughout data collection, study data collectors and the study coordinator will remain blinded to participants' exposure group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-low dietary sodium (Experimental): High sodium diet (3400 mg/day) feeding period followed by low sodium diet (2300 mg/day) feeding period
  Interventions: Other: High dietary sodium intake; Other: Low dietary sodium intake
- Low-high dietary sodium (Experimental): Low sodium diet (2300 mg/day) feeding period followed by high sodium diet (3400 mg/day) feeding period
  Interventions: Other: High dietary sodium intake; Other: Low dietary sodium intake

INTERVENTIONS:
Other: High dietary sodium intake — Fourteen day feeding period of high dietary sodium (3400 mg/day)
Other: Low dietary sodium intake — Fourteen day feeding period of low dietary sodium (2300 mg/day)

SUMMARY:
The overall objective of this study is to examine how dietary sodium is used by the body. In a racially diverse sample of adults, the investigators will examine the effects of high and low dietary sodium intake on the storage and excretion of sodium and determine whether sodium distribution affects blood pressure. This has implications for how investigators interpret studies that use urine biomarkers of sodium. Study findings about tissue sodium storage also have implications for managing hypertension and related conditions.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old;
* Diagnosed with high blood pressure or pre-hypertension (systolic blood pressure (SBP) > 120 mm Hg or diastolic blood pressure (DBP) > 80 mm Hg);
* Taking no more than two medications for high blood pressure;
* Currently has a primary care provider;
* Willing to eat all meals provided by the study for two 14-day feeding periods;
* Willing to complete study measurement procedures.

Exclusion Criteria:

* Diabetes;
* Smoker;
* Serious food allergies;
* Currently pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Estimated sodium concentration in skin and muscle | 60 days
  The concentration of sodium in skin and muscle will be measured, and the difference in concentrations resulting from high versus low sodium intakes will be calculated. Skin and muscle sodium stores will be non-invasively quantified using 23sodium-magnetic resonance imaging (23Na-MRI).
Estimated sodium concentration in bone | 60 days
  The concentration of sodium in bone will be measured, and the difference in concentrations resulting from high versus low sodium intakes will be calculated. Sodium storage in bone will be measured non-invasively using in vivo neutron activation analysis (IVNAA) technology to quantify the concentration of Na in the hand.
Concentration of sodium, potassium, and hormone regulators in excreted urine | 60 days
  Urinary concentration of sodium, potassium, and hormones (renin, angiotensin, aldosterone, free cortisol, free cortisone, glucocorticoid, and mineralocorticoid) will be measured and variation over time will be calculated.
Blood pressure | 60 days
  Blood pressure under high versus low dietary sodium conditions will be measured.

SECONDARY OUTCOMES:
Racial differences in concentrations of sodium in skin, muscle and bone | 60 days
  Blacks/African Americans mean sodium concentrations versus the average of the means of each of the other racial/ethnic groups will be examined.
Racial differences in concentration of urinary potassium excretion | 60 days
  The concentration of potassium excreted in urine will be compared between Blacks/African Americans versus the pooled sample of other racial/ethnic groups.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A Anderson, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States

DOCUMENTS (2):
  • Informed Consent Form: Main consent form (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT04110262/ICF_000.pdf
  • Informed Consent Form: Screening consent form (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT04110262/ICF_001.pdf